CLINICAL TRIAL: NCT02466594
Title: Impact of Active Thermoregulation on the Microcirculation of Free Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulf Dornseifer, MD (Other)
Responsible Party: Sponsor-Investigator, Ulf Dornseifer, MD, M.D., Klinik Bogenhausen
Organization: Klinik Bogenhausen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KBogenhausen
Record Dates: First submitted 2015-05-25; First posted 2015-06-09 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Microcirculation; Thermoregulation; Free Flap

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hilotherm Clinic® (Other): Intervention: Controlled Thermoregulation with Hilotherm Clinic® - Flap Temperature is altered by passive warming (dressing), active warming (38 C) and active cooling (10 C) each for 60 minutes following free flap transfer in every subject at the day of surgery and the following three days
  Interventions: Device: Hilotherm Clinic®

INTERVENTIONS:
Device: Hilotherm Clinic® — Controlled Thermoregulation using a water circulation based system (Hilotherm Clinic®). Controlled Thermoregulation with Hilotherm Clinic® - Flap Temperature is altered by passive warming (dressing), active warming (38 C) and active cooling (10 C) each for 60 minutes following free flap transfer in every subject at the day of surgery and the following three days

SUMMARY:
This study evaluates the impact of active thermoregulation on free flap microcirculation following free flap transfer. Thermoregulation is performed by passive warming, active warming (water circulation based device) and active cooling. Changes in microcirculation are assessed using combined laser Doppler flowmetry and remission spectroscopy.

DETAILED DESCRIPTION:
Measurements are conducted at the day of the operation as well as the first three days following the operation. Tissue temperature is assessed by a temperature measurement probe that is placed 8 mm underneath the skin. The microcirculation parameters of free perforator flaps are assessed using combined laser Doppler flowmetry and remission spectroscopy (O2C®). This allows non-invasive measurement of blood flow, capillary venous oxygen saturation and relative postcapillary filling pressure using a fiber optic probe that is placed on the flap surface. Controlled Thermoregulation (between 10 and 38°C) is enabled using a water circulation based system (Hilotherm Clinic®).

ELIGIBILITY:
Inclusion Criteria:

Patients receiving free perforator flaps with a skin island not less than 4x4 cm

Exclusion Criteria:

* non-compliance,
* non-consent,
* history of cardiac disease,
* arterial hypo- or hypertension,
* intake of vasoactive drugs,
* peripheral arterial occlusive disease,
* chronic kidney and liver disease,
* vasculitis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Blood Flow (AU) measured by Doppler flowmetry and remission spectroscopy (Oxygen to See, O2C®, Lea Medizintechnik, Giessen, Germany) | Measurements were conducted at the day of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Dornseifer, MD, Principal Investigator — Department of Plastic, Reconstructive, Hand and Burn Surgery, Bogenhausen Academic Hospital, Munich 81925, Germany
Locations (1):
- Department of Plastic, Reconstructive, Hand and Burn Surgery, Bogenhausen Academic Hospital, Munich 81925, Germany, Munich, Bavaria, Germany